CLINICAL TRIAL: NCT05646745
Title: Autologous Transobturator Fascia Lata Sling in Treatment of Female Stress Urinary Incontinence
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Mohamed Fawzy Abd Elfattah Salman, Director, Al-Azhar University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Fascia Lata TOT
Record Dates: First submitted 2022-12-03; First posted 2022-12-12 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Stress Urinary Incontinence
Keywords: Autologous; TOT; SUI; Stress
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Intervention Model Description: Autologous fascia lata is utilized via transobturator approach
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Autologous Fascia lata TOT (Experimental): Through incision in the lower lateral aspect of the thigh, 4 cm above the knee, ~1 cm× ~5 cm fascial strip is isolated from the fascia lata. Two stay sutures are secured to the corners of the fascial segment on each side.
  About 1cm skin incision is performed at the thigh fold on each side. Next, two separate trocar passages are performed on each side using a reusable C-shaped trocar, with care taken to ensure at least a 1 cm tissue bridge in the obturator membrane between the superior and inferior passes. Following this, the stay sutures are tied external to the obturator membrane on both sides, leaving the sling secured and flush with the mid-urethra. Sutures are also placed to secure the sling to the periurethral tissue to prevent rolling or migration of the fascial strip.
  Interventions: Procedure: Autologous Transobturator Fascia Lata Sling

INTERVENTIONS:
Procedure: Autologous Transobturator Fascia Lata Sling — Hydro-distention of the anterior vaginal wall, and a midline incision is made based on the mid-urethra. Dissection is carried out bilaterally to the obturator Foramen on both sides.
  Through incision in the lower lateral aspect of the thigh, 4 cm above the knee, ~1 cm× ~5 cm fascial strip is isolated from the fascia lata. Two stay sutures are secured to the corners of the fascial segment on each side.
  About 1cm skin incision is performed at the thigh fold on each side. Next, two separate trocar passages are performed on each side using a reusable C-shaped trocar, with care taken to ensure at least a 1 cm tissue bridge in the obturator membrane between the superior and inferior passes. Following this, the stay sutures are tied external to the obturator membrane on both sides, leaving the sling secured and flush with the mid-urethra. Sutures are also placed to secure the sling to the periurethral tissue to prevent rolling or migration of the fascial strip.

SUMMARY:
To evaluate the outcome of autologous transobturator fascia lata sling for treatment of female stress urinary incontinence at Al-Azhar university hospitals.

DETAILED DESCRIPTION:
Following induction of anesthesia and administration of perioperative antibiotics, the patient is positioned in the dorsal lithotomy position, sterilization and draping will be done. A sterile 16 French Foley catheter is placed to drain the bladder, following this, injectable normal saline is utilized using 10 cc syringe for hydro-distention of the anterior vaginal wall, and a midline incision is made based on the mid-urethra. Dissection is carried out bilaterally to the obturator Foramen on both sides.

Through incision in the lower lateral aspect of the thigh, 4 cm above the knee, ~1 cm× ~5 cm fascial strip is isolated from the fascia lata. Two stay sutures are secured to the corners of the fascial segment on each side.

About 1cm skin incision is performed at the thigh fold on each side. Next, two separate trocar passages are performed on each side using a reusable C-shaped trocar, with care taken to ensure at least a 1 cm tissue bridge in the obturator membrane between the superior and inferior passes. Following this, the stay sutures are tied external to the obturator membrane on both sides, leaving the sling secured and flush with the mid-urethra. Sutures are also placed to secure the sling to the periurethral tissue to prevent rolling or migration of the fascial strip.

ELIGIBILITY:
Inclusion Criteria:

* Women with genuine stress urinary incontinence.
* Mixed urinary incontinence with predominant stress element.
* Refractory cases to conservative therapy or patients who are not willing to consider (further) conservative treatment.

Exclusion Criteria:

* Mixed incontinence with predominant Urge urinary incontinence.
* Associated local abnormalities that may affect surgery outcomes (e.g. complete procidentia).
* Recent or active urinary tract infection.
* Recent pelvic surgery.
* Neurogenic lower urinary tract dysfunction.
* Previous surgery for stress urinary incontinence.
* Pregnancy
* Less than 12 months post-partum.
* Other gynaecologic pathologies affecting bladder functions ( eg, large fibroids, ovarian cysts)
* Genito-urinary malignancy.
* Current chemo or radiation therapy.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
complete cure | 3 months
  Number of patients without leakage with cough stress test and the patient is satisfied and on examination there is no leakage with cough test.

SECONDARY OUTCOMES:
improvement of SUI | 3 months
  Number of patients who report leakage only with severe exertion and using a smaller number of pads per day and she feels that she has improved. On examination there is no stress urinary incontinence.

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Mohamed Fawzy Salman, Cairo
  - Urology department - AlAzhar university, Cairo

IPD SHARING:
Plan to Share IPD: No